CLINICAL TRIAL: NCT03518775
Title: Repeatability and Reproducibility of the IOLMaster 700 Vers 1.70 and Agreement With IOLMaster 700 Vers. 1.50 and Pentacam
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Collaborators: ClinReg Consulting Services, Inc. (Other); Sierra Clinical Services, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: IOLMaster 2017-01909
Record Dates: First submitted 2018-04-06; First posted 2018-05-08 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Cornea
MeSH Terms: conditions — Corneal Diseases | interventions — Biometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Normal Eyes: Eyes with best-corrected visual acuity of 20/20 or better, and lens opacities of 1.0 or less in the study eye using the LOCS III system, and no prior Laser Vision Correction.
  Interventions: Device: Biometry
- Cataract Eyes: Cataract in the study eye greater than Grade 1 using the LOCS III system for one or more: nuclear opacity, nuclear color, cortical opacity, or PSC.
  Interventions: Device: Biometry
- Post LVC Eyes: History of Laser Vision Correction (LVC)
  Interventions: Device: Biometry

INTERVENTIONS:
Device: Biometry — Measurement of Cornea

SUMMARY:
The objectives of this study are to determine the agreement of measurements between the IOLMaster 700 SW Vers. 1.70 and IOLMaster 700 SW Vers. 1.50 and Pentacam, as well as to evaluate the repeatability and reproducibility of the IOLMaster 700 SW Vers 1.70.

The following parameters will be evaluated for Total Keratometry, (TK) and Posterior Corneal Surface (PCS):

* cylinder (CYL), Axis (A)
* spherical equivalent (SE)

Specific Objectives:

1. To compare the agreement of SE between IOLMaster 700 SW Vers. 1.70 and IOLMaster 700 SW Vers. 1.50 (Carl Zeiss Meditec AG, Jena, Germany)
2. To compare the agreement of Cylinder magnitude and axis between IOLMaster 700 SW Version 1.70 and Pentacam
3. To evaluate the repeatability and reproducibility of the IOLMaster 700 SW Vers. 1.70 for all measurement parameters listed above

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female 22 years of age and older.
2. No history of rigid contact lens wear for at least 2 weeks. Soft lenses, if worn, should be removed at least one hour prior to the measurement.
3. Able and willing to make the required study visits.
4. Able and willing to give consent and follow study instructions.
5. Group 1: normal eyes with best-corrected visual acuity of 20/20 or better, and lens opacities of 1.0 or less in the study eye using the LOCS III system, and no prior Laser Vision Correction.
6. Group 2: cataract in the study eye greater than Grade 1 using the LOCS III system for one or more: nuclear opacity, nuclear color, cortical opacity, or PSC.
7. Group 3: history of Laser Vision Correction (LVC).

Exclusion Criteria:

1. Previous intraocular surgery other than Laser Vision Correction in the study eye.
2. Previous corneal surgery other than Laser Vision Correction in the study eye.
3. Presence of any corneal or retinal abnormality on slit lamp examination in the study eye.
4. Corneal Cylinder < 0.75D measured with a IOLMaster.
5. Active ocular infection or inflammation.
6. Poor tear film/insufficient corneal reflex.
7. Best corrected visual acuity worse than 20/200 in the study eye.
8. Physical inability to be positioned at the slit-lamp biomicroscope or study devices (e.g. torticollis, head tremor, etc.).
9. Insufficient eyelid opening or eyelashes which partially conceal alignment or keratometry reflections and prevent capture of all measurements.
10. Inability to fixate (e.g. due to nystagmus, amblyopia or ocular disease, such as macular degeneration).
11. Rigid contact lens wear during past two weeks.
12. Principal Investigator's determination that the subject is not suitable due to other medical condition (reasons to be listed on eCRFs).

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be three cohorts: normal eyes (Group 1), cataract eyes (Group 2), and post Laser Vision Correction (LVC) eyes (Group 3), with no cross-over between the study groups.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Measurement Agreement between IOL Master Software Versions 1.70 and 1.50. | 1 hour
  IOLMaster 700 Vers. 1.70 SE_TK (Spherical Equivalent_Total Keratometry) Measurements will be compared to IOLMaster 700 SW Vers. 1.50 SE_K (Spherical Equivalent_Keratometry) Measurements for Agreement.
Measurement Agreement between IOLMaster Software Version 1.70 and Pentacam. | 1 hour
  IOLMaster 700 Vers. 1.70 A_TK (Axis_Total Keratometry), Cyl_TK (Cylinder_Total Keratometry), A_PCS (Axis_Posterior Corneal Surface), SE_PCS (Spherical Equivalent_Posterior Corneal Surface), and Cyl_PCS (Cylinder_Posterior Corneal Surface) Measurements will be compared to Pentacam Measurements for Agreement.
Repeatability and Reproducibility of IOLMaster 700 Software Version 700 Measurements. | 1 hour
  3. Evaluate the Repeatability and Reproducibility of the IOLMaster 700 SW Version 1.70 for A_TK, A_PCS, Cyl_TK, Cyl_PCS, SE_TK and SE_PCS.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Slade, MD, Principal Investigator — Slade & Baker Vision
Locations (1):
- Slade & Baker Vision, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogel A, Dick HB, Krummenauer F. Reproducibility of optical biometry using partial coherence interferometry : intraobserver and interobserver reliability. J Cataract Refract Surg. 2001 Dec;27(12):1961-8. doi: 10.1016/s0886-3350(01)01214-7. PMID 11738911
- [Background] Lu MJ, Zhong WH, Liu YX, Miao HZ, Li YC, Ji MH. Sample Size for Assessing Agreement between Two Methods of Measurement by Bland-Altman Method. Int J Biostat. 2016 Nov 1;12(2):/j/ijb.2016.12.issue-2/ijb-2015-0039/ijb-2015-0039.xml. doi: 10.1515/ijb-2015-0039. PMID 27838682
- [Background] Baumeister M, Terzi E, Ekici Y, Kohnen T. Comparison of manual and automated methods to determine horizontal corneal diameter. J Cataract Refract Surg. 2004 Feb;30(2):374-80. doi: 10.1016/j.jcrs.2003.06.004. PMID 15030827